CLINICAL TRIAL: NCT00248872
Title: A Randomized Trial of Changing Medication Adherence In Hypertensive African-American Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Mary E. Charlson, MD, Principal Investigator, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N01-HC-25196 (0203-704); N01HC25196 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: African-American; Hypertension; Medication adherence; Risk reduction
MeSH Terms: conditions — Hypertension; Medication Adherence; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): This group received follow-up every 2-months for one year. Follow-up included questions about their blood pressure and how well they had been able to adhere to their medication goal.
- Intervention Group (Experimental): This group received follow-up every 2-months for one year. Follow-up included questions about their blood pressure and how well they had been able to engage adhere to their medication goal. The intervention included receiving an additional educational workbook about using positive affect and self affirmation, as well as participating in using positive affect and self-affirmation to motivate behavior change, which in this case was to increase their physical activity level.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — During the physical activity goal setting process, subjects were randomly assigned to either the control or the intervention group. The intervention included receiving an additional educational workbook about using positive affect and self affirmation, as well as participating in using positive affect and self-affirmation to motivate behavior change, which in this case was to increase their medication adherence. Patient also received small token gifts to remind them of their participation in the study and to induce positive affect. The control group also set a physical activity goal and received the same follow-up, but did not participate in the positive affect and self-affirmation portion.
  Other Names: Positive affect and self-affirmation induction
  Arms: Intervention Group

SUMMARY:
The long-term objective is to determine whether better adherence to prescribed medications can be achieved through positive affect induction and self-affirmation leading to reduction in hypertension-related outcomes such as end-stage renal disease, stroke, and cardiovascular mortality among African American patients with poorly controlled hypertension.

DETAILED DESCRIPTION:
The objective of this randomized trial is to evaluate, among African American patients with poorly controlled hypertension, whether a novel intervention of positive affect induction and self-affirmation is more effective than usual care in increasing adherence to prescribed antihypertensive medications. The main outcome will be the change in medication adherence rate from enrollment to 12 months, which is defined as percentage (%) of prescribed doses taken by the patient during the interval of observation as measured by electronic medication event monitoring system (MEMS).

2. Secondary objectives

1. To determine, among African American patients with poorly controlled hypertension, the extent to which positive affect induction and self-affirmation influence patients' self-efficacy.
2. To determine, among African American patients with poorly controlled hypertension, the extent to which positive affect induction and self-affirmation influence medication adherence in those with significant depressive symptomatology (CES-D score > 16).
3. To determine, among African-American patients with poorly controlled hypertension, the extent to which positive affect induction and self-affirmation influence blood pressure control.
4. To explore the health beliefs of hypertensive African-American patients, regarding the meaning, causes and treatment of hypertension. In addition, the factors that facilitate and prevent adherence to prescribed antihypertensive medications will also be explored using a qualitative approach.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be self-identified as African-Americans.
2. All patients must be aged 18 years and older.
3. All patients must be diagnosed as having hypertension: For this project, hypertension will be defined according to the widely accepted criteria of the 6th Joint National Committee (JNC VI) Guidelines on Prevention, Detection, Evaluation and Treatment of Hypertension, which is a systolic blood pressure > 140 mm hg or a diastolic blood pressure > 90 mm hg or if participants are taking any prescribed antihypertensive medication.
4. Patients must be able to provide informed consent in English.

Exclusion Criteria:

1. Patients who are unable to walk several blocks for any reason.
2. Patients who refused to participate
3. Patients who are unable to provide informed consent.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2006-09 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Within patient change in medication adherence as measured by the MEMS cap. | Every two months for one year

CONTACTS AND LOCATIONS:
Overall Officials: Carla Boutin-Foster, MD,MS, Principal Investigator — Weill Medical College of Cornell University; Gbenga Ogedegbe, MD, MS, Principal Investigator — Columbia University; Mary E Charlson, MD, Study Director — Weill Medical College of Cornell University
Locations (1):
- The New York Presbyterian Hospital-Weill Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No Plan to Share IPD

REFERENCES:
- [Background] Boutin-Foster C, Ravenell JE, Greenfield VW, Medmim B, Ogedegbe G. Applying qualitative methods in developing a culturally tailored workbook for black patients with hypertension. Patient Educ Couns. 2009 Oct;77(1):144-7. doi: 10.1016/j.pec.2009.03.008. Epub 2009 Apr 16. PMID 19375264
- [Background] Boutin-Foster C, Ogedegbe G, Ravenell JE, Robbins L, Charlson ME. Ascribing meaning to hypertension: a qualitative study among African Americans with uncontrolled hypertension. Ethn Dis. 2007 Winter;17(1):29-34. PMID 17274206
- [Result] Ogedegbe GO, Boutin-Foster C, Wells MT, Allegrante JP, Isen AM, Jobe JB, Charlson ME. A randomized controlled trial of positive-affect intervention and medication adherence in hypertensive African Americans. Arch Intern Med. 2012 Feb 27;172(4):322-6. doi: 10.1001/archinternmed.2011.1307. Epub 2012 Jan 23. PMID 22269592